CLINICAL TRIAL: NCT00146783
Title: Efficacy of Sulphadoxine-pyrimethamine and Amodiaquine Alone or in Combination as Intermittent Preventive Treatment in Pregnancy in the Kassena-Nankana District of Ghana: a Randomized Controlled Trial
Brief Title: Navrongo Drug Options for IPT in Pregnancy Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Ministry of Health, Ghana (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: ITCR5096
Record Dates: First submitted 2005-09-05; First posted 2005-09-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Malaria
Keywords: intermittent preventive treatment; malaria; pregnancy; efficacy; safety
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Sulphadoxine-pyrimethamine
Drug: Sulphadoxine-pyrimethamine, amodiaquine

SUMMARY:
In areas of stable transmission, pregnant women, especially during the first and second pregnancies, have an increased susceptibility to Plasmodium falciparum malaria, malaria-related anaemia and an increased risk of having low birthweight babies. Intermittent Preventive Treatment in pregnancy(IPTp) with sulphadoxine-pyrimethamine has been shown to be effective in reducing the effects of malaria in pregnancy. This has mainly been in areas of perennial transmission and there is a need to study this effect in intense seasonal transmission settings. The emergence and spread of resistance to SP is likely to undermine its useful lifespan and it is important that other antimalarials that are safe and effective are identified for use in IPTp. The options are however limited. Amodiaquine has been shown to be effective in treatment of clinical cases of malaria, even in areas where chloroquine resistance is prevalent, and its combination with SP has been associated with favourable results. Both are affordable. However, there is limited data on their use in pregnancy. This study aims to assess the efficacy of SP in an area of intense seasonal transmission, and evaluate the safety and efficacy of amodiaquine and a combination of sulphadoxine-pyrimethamine and amodiaquine as possible alternatives to SP for use as IPTp.

DETAILED DESCRIPTION:
Background Pregnant women, particularly during the first and second pregnancy, have a high risk of Plasmodium falciparum infection and these infections are often asymptomatic but lead to maternal anaemia and low birth-weight. One approach to preventing malaria in pregnancy is prompt effective management of clinical malaria. In areas of moderate and high transmission however, peripheral parasitaemia is not a sensitive indicator as many women with placental parasitaemia may not have peripheral parasitaemia. Another option is to administer full curative doses of an effective antimalarial drug at predefined intervals during pregnancy (IPTp) without screening for parasitaemia. The efficacy of IPTp has been studied mostly in areas of high perennial transmission in Kenya and Malawi. IPTp has however been little investigated in West Africa where transmission is often intense and highly seasonal. It may not be appropriate to translate results between areas with different ranges of transmission intensities across the sub-Saharan African region and there is a need to study the effect of IPTp in highly seasonal intense transmission areas in West Africa.

IPTp with SP has been shown to be effective in reducing maternal anaemia, prevalence of placental parasitaemia and the incidence of low birth weight. SP offers a reasonable combination of ease of use and associated increased compliance, low cost, and relatively good tolerance and safety. However, the useful therapeutic life (UTL) predicted for SP is likely to be short, in part due to its prolonged half-life, causing a higher probability of selecting resistant strains and consequent rapid development of resistance. The emergence and spread of SP resistance will increasingly undermine this strategy, depleting the currently available and affordable drugs usable for intervention during pregnancy. It is therefore important that alternative antimalarials that are safe and effective in pregnancy are identified.

Specific primary objective To assess and compare the efficacy of a combination of sulphadoxine-pyrimethamine and amodiaquine, sulphadoxine-pyrimethamine or amodiaquine used as IPTp, in reducing the incidence of anaemia(Hb<11g/dl) at weeks 34-36 among primigravidae and secundigravidae.

Specific secondary objectives

To evaluate the effect of SP/AQ, SP or AQ on:

1. The mean birthweight of infants among primigravidae and secundigravidae
2. The incidence of clinical malaria during pregnancy among primigravidae and secundigravidae
3. The prevalence of anaemia (Hb <11g/dl) at delivery among primigravidae and secundigravidae
4. The prevalence of placental parasitaemia among women in their first or second pregnancies delivering at health facilities or by trained TBAs
5. The prevalence of peripheral parasitaemia at weeks 34-36 among primigravidae and secundigravidae
6. The prevalence of maternal peripheral parasitaemia at delivery among primigravidae and secundigravidae
7. To determine the safety and tolerability of AQ, SP used alone and in combination, among pregnant women of all parities
8. To determine the prevalence of molecular markers of resistance to AQ and SP among pregnant women who have malaria parasitaemia at enrolment
9. To document the factors that influence women's attitude towards ANC attendance, use of chemoprophylaxis and ITNs, and to determine what informs their choice to deliver at a particular facility

STUDY SITE The study will be carried out in the Kassena-Nankana district of northern Ghana. The residents are mainly subsistence farmers. There are two main seasons, a short wet season from June to September, during which the transmission of Plasmodium species peaks and a long dry season. The primary resource of the Navrongo Health Research Centre is a district-wide surveillance system, the Navrongo Demographic Surveillance System (NDSS), a longitudinal population registration system that is updated every 90 days. The district has 4 health centres, 3 clinics and a 140-bed hospital that serves as a referral centre. Information collated for the year 2002 in the Kassena-Nankana district indicated that out of an expected 6050 pregnancies, 95% registered for ANC, the average number of visits being 2.7. There were 2173(36%) supervised deliveries, 1279 of these at health facilities and 894 by trained TBAs. 794 out of 2405(33%) pregnant women had haemoglobin levels less than 10g/dl at registration.

STUDY POPULATION Pregnant women between 16 -32 weeks gestation attending antenatal care clinics at the district hospital or any of the four main health centres in the district will be eligible to join the study. The main endpoints will be assessed in primigravidae and secundigravidae however safety data will be collected for all women.

STUDY DESIGN The study will be carried out in two phases, a pre-intervention phase which will document women's knowledge, attitudes and practices on antenatal care, chemoprophylaxis and use of insecticide treated bednets and factors that influence their choice of where to deliver. The second phase, which is the intervention, will be a three-arm randomized blinded controlled trial.

Intervention study - Enrolment procedure The study will be explained to women as a group before each day's ANC activities begin. In order not to interfere with the routine ANC activities women who may want to be recruited will then proceed to the study team after their routine ANC care. After obtaining informed consent, socio-demographic information, an obstetric history including previous ANC attendances during current pregnancy, a history of any illness in the past week, and information on bed net use will be collected. Gestational age will be obtained from the ANC card as assessed by the midwife. Anthropometric indices measured will be weight, height and mid-upperarm circumference. The blood pressure and axillary temperature will also be measured. Fingerstick blood sample will be drawn for haemoglobin testing, malaria thick blood smear and filter paper samples, after which each woman will be assessed for eligibility. Subjects will be randomized individually to receive the study drugs. The code on the envelope will be written on all the study forms and samples. The subject's name, address and date of first dosing will be noted on the envelope, to ensure that each woman receives the right regimen over the three-day period and also during subsequent doses of IPTp. To ensure compliance, all doses will be supervised either at the health facility, or through home visits (on Days 1 and 2). Women will receive between one and three doses of the drugs, depending on gestational age at recruitment, thus women recruited at 16 - 19 weeks will receive three doses, those recruited at 20 -26 weeks, two doses and those recruited from 27 -32weeks, one dose. The interval between dosing schedules will be 8 weeks, however the minimum interval allowed will be 4 weeks.

All women will be encouraged to deliver at a health facility or by a trained traditional birth attendant, and they will be given an identification card to take to the health facility so that the necessary samples can be taken and labelled adequately during delivery. These identification cards will also bear a note that the woman may have received AQ, SP or a combination as IPTp and should therefore not be given those drugs for clinical malaria, to avoid women being given repetitive doses within short intervals of time. Such women will be given Quinine 10mg/kg 8 hourly for 7days as recommended by the national treatment guidelines.

Assessment of drug tolerance and adverse drug reactions All women will be visited at home between Days 7 and 10 to look for any adverse events due to the study drugs. They will be advised to report to a health facility if they should experience any untoward effect of the drugs prior to, or after this home visit. The frequency and severity of spontaneous and elicited adverse events will be recorded. In the light of the information obtained, the association between the event and any of the study drugs will be judged as per the WHO guidelines52. All serious and adverse events will be reported to the DSMB immediately, and followed up with a written report which will fully document the event, and any available laboratory information or clinical data, will be included in the report.

Follow-up At subsequent visits for IPTp and at weeks 34 -36, a simple questionnaire will be administered to assess the presence of malaria symptoms, potential side effects of the study drugs since the last assessment, and bednet use. To ensure that women complete subsequent doses of IPTp, lists of women due for second or third doses will be computer-generated, and they will be reminded at least a week before the next dose is due to attend the ANC. At 34 -36 weeks blood samples will be taken to assess for haemoglobin levels (Hb) and peripheral parasitaemia. Women with severe anaemia (Hb levels <7g/dl) will be referred to the hospital for further investigations and management. Women who do not turn up at the ANC will be followed up at home to collect the blood sample. Blood slides from symptomatic women will be read immediately and women found to have parasitaemia will be given Quinine 10mg/kg 8 hourly for 7 days as per national treatment guidelines.

Delivery Women delivering at the hospital will have bloodsmears made from a fingerprick, and maternal side of the placenta, and have Hb level assessed. Women delivering at the health centre will have placental blood smears, and a peripheral blood smear taken. Those delivered by TBAs will have the placental smear taken.

Blood samples for haemoglobin estimation for women delivering at the health centre or by TBAs will be taken at home within 7 days of delivery. Assessment of Hb will be carried out on women who delivered spontaneously without any complications such as post-partum haemorrhage at the hospital on day of delivery to 7days post delivery, to construct a nomogram which would be used to estimate the haemoglobin levels at delivery for women who delivered at the health centre or by TBA who could not have an Hb done on day of delivery for logistic reasons.

All infants delivered at the hospital or health centre will be weighed and gestational age assessed by a modification of Dubowitz's examination within 24 hours of delivery53. To ensure that birthweights of infants delivered at home are taken within seven days of delivery, a list of women with gestation of 34 weeks or more will be generated according to area of residence. This would be given to Community Key Informants (CKI) who would be contacted weekly by field staff for information on those who were delivered by TBAs or at home. A follow-up will then be made to take the weight of the babies. Mothers will be encouraged to inform CKIs soon after delivery. The TBAs will be asked to inform CKIs whenever they delivered a study subject, so that the samples can be collected.

Infants for whom the Dubowitz score is obtained will be classified as follows:

Premature -LBW : gestational age is <37weeks and birthweight is <2500g IUGR-LBW: gestational age is ≥ 37weeks and birthweight is <2500g Normal birthweight : birthweight is ≥ 2500g

Withdrawal from study A withdrawal shall be any enrolled subject who does not complete the study as planned. This may be due to (a) withdrawal of consent, (b) reaction attributable to any of the study drugs or (c) termination of pregnancy (abortions or miscarriages). A withdrawal form shall be filled for such persons, indicating reasons for withdrawal, and they will be followed up for outcome measures, unless they decline to give consent.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with gestation between 18-32weeks,
* willing to give written consent to take part in the study
* Resident in the study area and available for follow-up.

Exclusion Criteria:

* Presentation with clinical symptoms of malaria (this would not affect subsequent enrollment at a later date),
* Known allergies or reactions to study drugs,
* Medical conditions needing hospital admission.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3642 (Actual)
Dates: Start 2004-06; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
HB at delivery | with inseven 7days of delivery

SECONDARY OUTCOMES:
placental malaria | on the day of delivery
maternal peripheral parasitaemia at delivery | within seven days of dellivery
tolerance and adverse events after taking study drugs
molecular markers of drug resistance to SP and Amodiaquine

CONTACTS AND LOCATIONS:
Overall Officials: Christine Clerk, MBChB, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Daniel Chandramohan, MBBS, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Brian Greenwood, FRCP, FRS, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Navrongo District Hosptial, Navrongo, Upper East Region, Ghana

REFERENCES:
- [Derived] Clerk CA, Bruce J, Affipunguh PK, Mensah N, Hodgson A, Greenwood B, Chandramohan D. A randomized, controlled trial of intermittent preventive treatment with sulfadoxine-pyrimethamine, amodiaquine, or the combination in pregnant women in Ghana. J Infect Dis. 2008 Oct 15;198(8):1202-11. doi: 10.1086/591944. PMID 18752443